CLINICAL TRIAL: NCT04332159
Title: Inhaled Methoxyflurane for Pain Management in Nasal Bone Fracture Reduction : A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Inhaled Methoxyflurane for Pain Management in Nasal Bone Fracture Reduction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Pierre-Hugues Fortier, M.D., Clinical professor, Otolaryngology and Head & Neck Surgery, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CÉR 2020-3355
Record Dates: First submitted 2020-01-27; First posted 2020-04-02 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Pain, Acute; Nasal Fracture
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: To reach their objectives, the investigators propose a randomized, double-blind, placebo-controlled study on a sample of patients randomized in two different groups:
  * Group A (intervention) : Closed nasal fracture reduction under local anesthesia and inhaled Methoxyflurane.
  * Group B (control) : Closed nasal fracture reduction under local anesthesia and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo in this study is a 0,9% saline solution that comes in an identical inhaler as the Methoxyflurane. The inhaler for both group will be prepared by the research pharmacist right before the procedure. The characteristic smell of the Methoxyflurane solution will be reproduced by pouring a few drops of Methoxyflurane just above the tip of the inhaler a couple of minutes before the administration of the Methoxyflurane or placebo (will be done for both groups by a pharmacy technician experienced in double-blind research - CIUSSS de l'Estrie-CHUS site Hôtel-Dieu) to make sure that the double-blind design is respected. The pharmacy is located inside the hospital near the outpatient clinic so packages will be easily available within minutes when patients are recruited. In addition, to lower the risk of group identification, a N-95 mask will be worn during each procedure by the investigators and the research nurse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Inhalation of Methoxyflurane through a Penthrox inhaler
  Interventions: Procedure: Closed nasal fracture reduction
- Control group (Placebo Comparator): Inhalation of placebo (0.9% salin solution) through a Penthrox inhaler
  Interventions: Procedure: Closed nasal fracture reduction

INTERVENTIONS:
Procedure: Closed nasal fracture reduction — Closed nasal fracture reduction is performed under local anesthesia with addition of Methoxyflurane or placebo

SUMMARY:
This is a randomised, double-blind, placebo controlled study to evaluate the efficacy of Methoxyflurane (Penthrox®) for the treatment of acute pain during closed nasal fracture reduction.

The study aims to provide evidence under blinded controlled conditions that Penthrox is safe and effective in patients aged 18 to 65 years during closed nasal fracture reduction.

DETAILED DESCRIPTION:
The main objective of this study is to establish if the addition of Methoxyflurane to local anesthesia has the ability to significantly reduce the pain during closed nasal fracture reduction compared to local anesthesia with placebo.

The secondary outcomes consist of assessing if inclusion of Methoxyflurane will have a positive impact on the time needed to achieve the reduction, the need for backup analgesia, the rate of reduction failure, pain level during infiltration of local anesthesia and the clinician's appreciation of the procedure.

As an hypothesis, the investigators expect that the addition of Methoxyflurane to the standard local anesthesia will significantly reduce the pain compared to local anesthesia with placebo during closed nasal fracture reduction. The investigators also think that Methoxyflurane might reduce the duration of the reduction, limit the need for backup analgesia, reduce the rate of reduction failure, reduce the pain level due to infiltration of local anesthesia and facilitate the procedure for the clinician.

To reach these objectives, the investigators propose a randomized, double-blind, placebo-controlled study on a sample of patients randomized in two different groups:

* Group A (intervention) : Closed nasal fracture reduction under local anesthesia and inhaled Methoxyflurane.
* Group B (control) : Closed nasal fracture reduction under local anesthesia and placebo.

The placebo in this study is a 0,9% saline solution that will come in an identical Penthrox inhaler. The inhaler will be prepared by a pharmacy technician experienced in double-blind research right before its use. The characteristic smell of the Methoxyflurane solution will be reproduced by pouring a few drops of Methoxyflurane just above the tip of the inhaler. N95 masks will be worn by the clinician and research nurse throughout the procedure to lower the risk of group identification.

PROCEDURE Patient referred to the investigators outpatient clinic for nasal fracture 7 to 10 days from the trauma date will be evaluated by one of the investigator and the need for intervention will be established.

Eligible patients will be randomised in a 1:1 ratio to have 17 patients per treatment arm (an interim analysis will be done after 10 patients per treatment arm). Eligible patients will receive either methoxyflurane or placebo from the PENTHROX® inhaler in a 1:1 ratio.

Before the procedure, the patient will assess his current level of pain on the visual analog scale (baseline pain). The patient will then self-administer 6 to 10 successive inhalations of Penthrox or placebo (assisted by the research nurse). The clinician will then wait 5 minutes before proceeding with local anesthesia as follow :

1. Two sprays of 4% lidocaine in each nostril.
2. Bilateral infratrochlear block with local 2% lidocaine with epinephrine 1:100000 (approximately 0.5 cc on each side). This will be done carefully to ensure that anatomical landmarks are preserved in order to obtain a proper reduction. (Infiltration of the skin on the lateral walls of the nose right above the proper nasal bone)
3. Bilateral infra-orbital block through the buccal mucosa using local 2% lidocaine with epinephrine 1:100 000 (approximately 1.5 cc on each side)
4. Efficacy of the local lidocaine is evaluated and additional infiltration will be done when needed.
5. Packing of the nose with cotton balls soaked with 10 cc of a ½ lidocaine- ½ oxymetazoline solution. (4% lidocaine)

The patient will use the inhaler one more after local anesthesia and the investigator will wait 5 minutes prior to proceeding with the closed reduction to ensure an adequate efficacy of the topical lidocaine-oxymetazoline anesthesia.

The cotton balls will then be removed and the clinician will proceed with the closed reduction.

The research nurse then documents the time at which the reduction begins. A scalpel handle is placed against the external nose to measure the distance from the medial canthus to the nostril rim. The scalpel handle is inserted between the depressed nasal bone and the the nasal septum, parallel to the nasal dorsum. The depressed bone is pulled laterally and guided into a neutral position with the scalpel handle while direct pressure is applied medially on the contralateral nasal bone (the laterally deviated side) in order to push it back into its neutral position. If needed, centrally depressed fragments require an anterior lifting motion with the elevator. These steps are repeated until the patient and the clinician are satisfied with the aesthetic result or if the patient asks the clinician to stop the procedure. End time of the procedure will also be noted.

The patient can ask for additional Methoxyflurane inhalations at anytime during the procedure. The patient is provided with 3 mL bottle of Methoxyflurane (or placebo) and cannot ask for another one. If during the procedure the patient asks for additional analgesia, his nose will be packed with cotton balls soaked in lidocaine-oxymetazoline for 5 minutes. However, if despite additional analgesia the procedure is interrupted because it is too painful for the patient, it will be considered as a reduction failure due to pain (whether the procedure is carried out under systemic analgesia, sedation or is abandoned). In the event of failure to achieve adequate fracture reduction, sedation and/or general anesthesia will be offered to the patient to complete the reduction.

After the procedure, pain levels (during infiltration of local anesthesia, mean and peak pain during the reduction) will be reported on the visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Being a man or a woman between 18 and 75 years old, inclusively ; and
* Being covered by the Quebec medical insurance (RAMQ); and
* Presenting an uncomplicated nasal fracture requiring a delayed (7 to 10 days) closed reduction.

Exclusion Criteria:

* Pregnant or breastfeeding woman; or
* Known for renal insufficiency (DFG < 50) ; or
* Known for hepatic impairment; or
* Personal or familial allergies/hypersensitivity to fluorinated products; or
* Contraindications to local anesthesia (including allergies); or
* Personal or family history of malignant hyperthermia; or
* Other facial fractures and/or significant injuries; or
* Altered state of consciousness (dementia, drug intoxication, head trauma or other similar psychologic disorder); or
* Significant respiratory impairment; or
* Haemodynamic instability; or
* Simultaneous use of alcohol, isoniazid, phenobarbital, rifampin, opioids, sedatives, hypnotics, sedative antihistaminics, general anesthetics, phenothiazines, tranquilizers, myorelaxants, nephrotoxic antibiotics (tetracycline, gentamicin, colistine, polymyxin B, amphotericin B); or
* Use of cannabis or other illicit drugs the day of the procedure; or
* Use of pain medication in past 6 hours; or
* Use of Methoxyflurane : more than 6 mL in the last 48 hours or more than 15 mL in the last week or usage in the last 3 months; or
* Need of sedation or general anesthesia for the procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain level variation during nasal closed reduction: visual analog scale | The "baseline pain" will be assessed before local anesthesia will be administered (at the very beginning of the procedure), whereas the "mean pain" and the "peak pain" will be assessed after the closed reduction is completed.
  The primary outcome is pain level variation during the closed reduction. Three pain levels will be collected using the visual analog scale :
  * Pain level before the procedure (or "baseline pain") : will be assessed in order to analyse pain variation during the procedure between the two groups
  * Mean pain level during the procedure (or "mean pain"), defined as the average amount of pain felt throughout the procedure by the patient
  * Peak pain level during the procedure (or "peak pain"), defined as the worst pain that the patient had felt during the procedure
  The visual analog scale is a validated scale on which patients are asked to report their pain level, from zero (absence of pain) to 10 (worst pain imaginable).
  Pain variation during the procedure will be assessed using two outcome measures :
  1. The mean pain due to procedure (the difference between the "mean pain" and the "baseline pain")
  2. The peak pain during the procedure, as measured on the visual analog scale

SECONDARY OUTCOMES:
Time needed to achieve the reduction | The time needed to achieve the reduction will be calculated by subtracting the time at the beginning of the reduction to the time at the end of the reduction, which will be documented by a research nurse during the procedure.
  Time needed to achieve closed reduction, from the beginning of the reduction manoeuvres until nasal reduction is completed, will be monitored and compared between the two groups. (This will not take into account the time taken for Methoxyflurane administration and local anesthesia infiltration.)
Rate of participants requesting backup analgesia during the procedure | Immediately after the intervention
  The need for additional analgesia during the procedure will be documented and compared between the two groups, more precisely
  1. Additional use of inhaler
  2. Lidocaine-oxymetazoline cotton balls At the end of the procedure, the investigator will document if the patient requested backup analgesia during the procedure.
Reduction failure rate | Immediately after the intervention
  Reduction failure due to inadequate pain management despite additional measures will be documented and compared between the two groups
Pain level during anesthesia: visual analog scale | Immediately after the intervention
  Pain level during infiltration of local anesthesia will be assessed on a visual analog scale and compared between the two groups
  The visual analog scale is a validated scale on which patients are asked to report their pain level, from zero (absence of pain) to 10 (worst pain imaginable).
Number of procedures limited by pain | Immediately after the intervention
  After the procedure, the investigator will assess, by answering "yes" or "no", If he believed that the pain felt by the participant was limiting the execution of the closed nasal reduction and therefore jeopardizing the aesthetic result

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No